CLINICAL TRIAL: NCT06225492
Title: Use of DaxibotulinimtoxinA Injection for Platysma Bands of the Neck
Brief Title: DaxibotulinimtoxinA for Treatment of Platysmal Neck Bands
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Main Line Center for Laser Surgery (Other)
Responsible Party: Principal Investigator, Kachiu Lee, MD, Physician, Main Line Center for Laser Surgery
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DAXI0823
Record Dates: First submitted 2024-01-09; First posted 2024-01-26 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Aging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- DaxibotulinumtoxinA 20 units (Experimental): Subjects will receive 20 units of daxibotulinumtoxinA per platysmal band, up to 2 anterior bands and 2 lateral bands.
  Interventions: Drug: DaxibotulinumtoxinA 20 units
- DaxibotulinumtoxinA 15 units (Experimental): Subjects will receive 15 units of daxibotulinumtoxinA per platysmal band, up to 2 anterior bands and 2 lateral bands.
  Interventions: Drug: DaxibotulinumtoxinA 15 units

INTERVENTIONS:
Drug: DaxibotulinumtoxinA 15 units — Subjects will be treated with 15 units of daxibotulinumtoxinA per platysmal band
  Other Names: Daxxify
  Arms: DaxibotulinumtoxinA 15 units
Drug: DaxibotulinumtoxinA 20 units — Subjects will be treated with 20 units of daxibotulinumtoxinA per platysmal band
  Other Names: Daxxify
  Arms: DaxibotulinumtoxinA 20 units

SUMMARY:
This study seeks to evaluate the effectiveness and duration of action of DaxibotulinumtoxinA for neck rejuvenation through treatment of platysmal bands. This study will consist of one treatment visit with subjects being randomized to receiving 15 or 20 units of DaxibotulinumtoxinA per platysmal band. Subjects will return for 5 follow-up visits at 8, 12, 16, 20, and 24 weeks for evaluation.

DETAILED DESCRIPTION:
This clinical investigation is a prospective study consisting of a screening/treatment visit and 5 follow-up visits. A total of 20 patients will be recruited.

Following informed consent and screening, each eligible subject will be photographed. Next, patients will be randomized to receive 15 or 20 units of DaxibotulinumtoxinA per platysmal band. Patients randomized to each group will receive the same dosage injected to each neck band divided over 4 to 5 injection sites (up to 2 anterior and 2 lateral platysmal bands).

After randomization, patients will be treated with either 15 or 20 units per band. After treatment, subjects will be provided with post treatment instructions. Randomization will be conducted by having the patient pick either "15" or "20" out of a box. A total of 10 patients will be randomized to the 15 unit/platysmal band group. Another 10 patients will be randomized to the 20 unit/platysmal band group. The physician will fill out the 5-point Merz Neck Scale at baseline and at each follow-up visit. Photographs will be captured at each visit.

The patient will return at post-treatment weeks 8, 12, 16, 20, and 24. Subjects will fill out FACE-Q Satisfaction with Outcome surveys at each follow-up visit. FACE-Q Appraisal of Neck surveys will be filled out by the patient at the baseline and follow-up visits.

A blinded independent evaluator will evaluate the baseline and post-treatment photographs on Merz Neck Scale after completion of the study.

ELIGIBILITY:
Inclusion Criteria:

* >30 years old
* Rating of 2, 3, or 4 on 5-point Merz Neck Scale
* No use of any botulinum toxin in the neck for the past 6 months

Exclusion Criteria:

* Pregnancy
* Prior adverse reaction or known hypersensitivity to neuromodulators treatment
* Connective tissue disorder
* Scar in the treatment area
* History of dysphagia and/or neuromuscular disorders (such as but not limited to Amyotrophic Lateral Sclerosis, Multiple sclerosis, Myasthenia Gravis, Lambert-Eaton syndrome, others per PI's discretion)
* Active infection in treatment area
* Active moderate or severe inflammatory disease in treatment area such as atopic dermatitis, psoriasis
* Prior treatment with neuromodulators in treatment area (neck) within the past 6 months

Min Age: 31 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Effectiveness of DaxibotulinumtoxinA for platysmal neck bands measured on Platysmal Neck Banding Scale | 3 months
  Platysmal Neck Banding Scale (Scored on a 0-4 scale with 4 being the most severe)

SECONDARY OUTCOMES:
Evaluate patient-reported outcomes (patient satisfaction with neck using FACE-Q scale) | 3 months
  Patient satisfaction with neck using FACE-Q scale (scored on a 1-100 scale with 100 being highest satisfaction)

CONTACTS AND LOCATIONS:
Overall Officials: Kachiu Lee, MD, Principal Investigator — Physician
Locations (1):
- Main Line Center for Laser Surgery, Ardmore, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Final data from study is available to share upon request.
Supporting Information: Study Protocol, SAP
Time Frame: 5 years
Access Criteria: IRB approval